CLINICAL TRIAL: NCT02124018
Title: Post Myocardial Infarction Risk Stratification for Sudden Cardiac Death in Patients With Preserved Ejection Fraction: PRESERVE-EF
Brief Title: Risk Stratification in Patients With Preserved Ejection Fraction
Acronym: PRESERVE-EF
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: Medtronic (Industry); General Electric (Industry)
Responsible Party: Principal Investigator, Kostantinos A. Gatzoulis, Assoc. Professor of Cardiology, University of Athens
Other Study IDs: UOA-PRESERVE1
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Risk stratification; Sudden cardiac death; Preserved ejection fraction; Programmed ventricular stimulation
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post-MI patients: Asymptomatic post-MI patients late after MI or 40 days after STEMI-NSTEMI with preserved ejection fraction and absence of active ischemia Programmed ventricular stimulation (PVS) will be performed in high-risk patients based on non-invasive evaluation.
  ICD implantation will be performed in patients with induced ventricular tachycardia (VT) upon PVS
  Interventions: Procedure: Programmed ventricular stimulation; Device: ICD implantation

INTERVENTIONS:
Procedure: Programmed ventricular stimulation — Programmed ventricular stimulation in high-risk patients based on non-invasive evaluation
Device: ICD implantation — ICD implantation in patients with induced VT in programmed ventricular stimulation

SUMMARY:
The purpose of the study is to assess the prevalence and the prognostic value of non-invasive indexes and programmed ventricular stimulation for sudden cardiac death in post-myocardial infarction (MI) patients with left ventricular ejection fraction (LVEF)>40%.

DETAILED DESCRIPTION:
1000 asymptomatic post-MI patients>40%, at least 40 days post-MI, revascularized or without needing further revascularization (in any case without any evidence of ischemia) will be enrolled.

The patients will be divided into two categories:

1. Asymptomatic patients with revascularized ST-elevation MI (STEMI) (remaining stenoses in non culprit vessels <70%) at 40 days post-MI (when LVEF>40% will be re-assessed)
2. Asymptomatic patients late (at any time after 40 days) after MI (initially STEMI-NSTEMI at discharge Q-non Q) with LVEF>40% right after a negative stress test or right after a negative for stenoses control coronary catheterization All patients will undergo non-invasive evaluation (ECG, Holter monitoring and 45-min high resolution recording). In case they fulfill at least one out of seven pre-specified criteria they will undergo programmed ventricular stimulation and implantable cardioverter-defibrillator (ICD) implantation (if inducible) All patients will be followed-up for 3 years for sudden cardiac death and its surrogate (appropriate ICD activation)

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients with revascularized STEMI (remaining stenoses in non culprit vessels <70%) at 40 days post-MI (when LVEF>40% will be re-assessed)
* Asymptomatic patients late after MI (initially STEMI-NSTEMI at discharge Q-non Q) with LVEF>40% right after a negative stress test or right after a negative for stenoses control coronary catheterization

Exclusion Criteria:

* Episodes of sustained VT or aborted sudden cardiac death (SCD) 48 hours after the acute MI phase.
* Episodes of syncope within the last 6 months
* Cancer, liver failure (cirrhosis), end-stage renal disease
* Use of anti-arrhythmic drugs other than b-blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 asymptomatic post-MI patients>40%, at least 40 days post-MI, revascularized or without needing further revascularization (in any case without any evidence of ischemia)
  The patients will be divided into two categories:
  1. Asymptomatic patients with revascularized STEMI (remaining stenoses in non culprit vessels <70%) at 40 days post-MI (when LVEF>40% will be re-assessed)
  2. Asymptomatic patients late after MI (initially STEMI-NSTEMI at discharge Q-non Q) with LVEF>40% right after a negative stress test or right after a negative for stenoses control coronary catheterization
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gatzoulis, MD, PhD, Principal Investigator — University of Athens, Hippokration Hospital
Locations (1):
- First Cardiology Clinic, Hippokration Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gatzoulis KA, Tsiachris D, Arsenos P, Antoniou CK, Dilaveris P, Sideris S, Kanoupakis E, Simantirakis E, Korantzopoulos P, Goudevenos I, Flevari P, Iliodromitis E, Sideris A, Vassilikos V, Fragakis N, Trachanas K, Vernardos M, Konstantinou I, Tsimos K, Xenogiannis I, Vlachos K, Saplaouras A, Triantafyllou K, Kallikazaros I, Tousoulis D. Arrhythmic risk stratification in post-myocardial infarction patients with preserved ejection fraction: the PRESERVE EF study. Eur Heart J. 2019 Sep 14;40(35):2940-2949. doi: 10.1093/eurheartj/ehz260. PMID 31049557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2014 to July 2018, 575 consecutive patients were enrolled in the seven Departments of Cardiology participating in the study
Groups:
- Low Risk Group: No Non-Invasive Risk Factors (NIRFs) present - no invasive programmed ventricular stimulation (PVS) performed
- Intermediate Risk Group: At least one NIRF present - noninducible upon programmed ventricular stimulation (PVS) (no sustained ventricular tachyarrhythmia was induced i.e. either with a duration >30seconds or causing hemodynamic instability necessitating termination)
- High Risk Group: At least one NIRF present AND inducible upon PVS (sustained ventricular tachyarrhythmia was induced).
Period: Overall Study
Arm/Group | Low Risk Group | Intermediate Risk Group | High Risk Group
Started | 371 | 111 | 41
Completed | 371 | 111 | 41 (Numbers do not add up to 575 (enrolled) due to refusals of programmed ventricular stimulation)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to some patients' refusal to be submitted to invasive programmed ventricular stimulation, 52 patients were unstratifiable (unknown if Group 2 or 3), and thus 371+111+41=523=575-52
Groups:
- Low Risk Group: No NIRFs present - no invasive PVS performed
- Intermediate Risk Group: At least one NIRF present - noninducible upon PVS
- High Risk Group: At least one NIRF present AND inducible upon PVS
- Total: Total of all reporting groups
Arm/Group | Low Risk Group | Intermediate Risk Group | High Risk Group | Total
Number analyzed (Participants) | 371 | 111 | 41 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.2) | 60 (10.9) | 61.7 (9.2) | 57 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 15 | 1 | 73
  Male | 314 | 96 | 40 | 450
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Greece | 371 | 111 | 41 | 523

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Arrhythmic Events (MAEs) - Present When One of the Following Occurred: Sudden Cardiac Death, Sustained Ventricular Tachycardia, or Implantable Cardioverter - Defibrillator (ICD) Activation
Description: The number of patients from each risk level group meeting the primary endpoint will be used to assess diagnostic accuracy (positive/negative predictive value, sensitivity and specificity) of the proposed two-stage, PVS-inclusive, risk stratification approach for the allocation of an ICD
Time Frame: From stratification completion (i.e. allocation to one of three risk level groups) until either occurrence of primary endpoint or study completion (mean 32months) - study stopped early due to emergence of clearly defined high risk subgroup
Measure: Number; unit: participants
Arm/Group | Low Risk Group | Intermediate Risk Group | High Risk Group
Number analyzed (Participants) | 371 | 111 | 41
participants | 0 | 0 | 9

2. Secondary Outcome: Total Mortality
Description: All-cause mortality
Time Frame: From completion of risk stratification to study completion or outcome occurrence (mean 32 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Group | Intermediate Risk Group | High Risk Group
Number analyzed (Participants) | 371 | 111 | 41
Participants | 0 | 4 | 1

ADVERSE EVENTS:
Time Frame: From stratification completion (allocation to one of risk level groups) to adverse event occurrence, or study completion - mean 32 months
Description: Adverse events due to PVS and ICD implantation
Arm/Group | Low Risk Group | Intermediate Risk Group | High Risk Group
All-Cause Mortality (participants affected / at risk) | 0/371 | 4/111 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/371 | 0/111 | 0/41
Other Adverse Events (participants affected / at risk) | 0/371 | 0/111 | 0/41

LIMITATIONS AND CAVEATS:
Study was not a randomized clinical trial since almost all patients with a per protocol indication received a device, without the presence of a high-risk control group, thus potentially overestimating true arrhythmic risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02124018/Prot_SAP_000.pdf